CLINICAL TRIAL: NCT04658589
Title: A Multicenter Prospective Phase II Comparative Study of Laparoscopic Versus Open Distal Gastrectomy After Neoadjuvant Chemotherapy for the Treatment of Locally Advanced Gastric Cancer Patients
Brief Title: Laparoscopic vs. Open Distal Gastrectomy After Neoadjuvant Chemotherapy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chonnam National University Hospital (Other)
Responsible Party: Principal Investigator, Young Kyu Park, Professor, Chonnam National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H2020-0407
Record Dates: First submitted 2020-12-01; First posted 2020-12-08 (Actual); Last update posted 2020-12-08 (Actual); Status verified 2020-12

CONDITIONS: Stomach Neoplasm
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laparoscopic distal gastrectomy (Experimental): Laparoscopic distal gastrectomy after neoadjuvant chemotherapy for the treatment of locally advanced gastric cancer patients
  Interventions: Procedure: Laparoscopic versus open distal gastrectomy
- Open distal gastrectomy (Active Comparator): Open distal gastrectomy after neoadjuvant chemotherapy for the treatment of locally advanced gastric cancer patients
  Interventions: Procedure: Laparoscopic versus open distal gastrectomy

INTERVENTIONS:
Procedure: Laparoscopic versus open distal gastrectomy — Laparoscopic versus open distal gastrectomy after neoadjuvant chemotherapy for locally advanced gastric cancer

SUMMARY:
The study was designed as single-country, multi-center, open-labelled, randomized (1:1), phase II trial.

238 patients with medically and technically operable advanced gastric adenocarcinoma in middle or distal 1/3 of stomach are enrolled and randomly assigned to laparoscopic gastrectomy group and open gastrectomy group. 4 cycles of mFLOT chemotherapy will be conducted before and after gastrectomy.

The primary objective of this study is comparison of D2 lymph node dissection compliance rate between open surgery group and laparoscopic surgery group after neoadjuvant chemotherapy.

DETAILED DESCRIPTION:
The effect of neoadjuvant chemotherapy on locally advanced gastric cancer was confirmed from a prospective clinical trial. Oncologic safety and excellence of the laparoscopic gastrectomy surgery was recently established for locally advanced gastric cancer.

However, neither technical nor oncologic stability was established for laparoscopic gastrectomy surgery after neoadjuvant chemotherapy. Anticipated benefits from laparoscopic gastrectomy surgery after neoadjuvant chemotherapy are as follows: 1) Reduced postoperative complications; 2) Reduced intra- or postoperative transfusion and patient's pain after surgery; 3) Enhance postoperative recovery (shortened hospitalization duration); 4) Facilitate completion rate of adjuvant chemotherapy.

The study was designed as single-country, multi-center, open-labelled, randomized (1:1), phase II trial.

238 patients with medically and technically operable advanced gastric adenocarcinoma in middle or distal 1/3 of stomach are enrolled and randomly assigned to laparoscopic gastrectomy group and open gastrectomy group. 4 cycles of mFLOT chemotherapy will be conducted before and after gastrectomy.

The primary objective of this study is comparison of D2 lymph node dissection compliance rate between open surgery group and laparoscopic surgery group after neoadjuvant chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who voluntarily expressed their consent to participate in this trial by signing a written 'Subject Consent Form.'
2. Patients whose gastric adenocarcinoma located in the middle or lower part of the stomach is histologically confirmed and deemed possible to perform a radical distal gastrectomy surgery.
3. Patients who come under T2/N(+)M0, T3~4a/N(- or +) M0 according to the 8th edition of the TNM classification.

Exclusion Criteria:

* Methodologies

  1. Patients less than 20 years old or older than 80 years old
  2. Eastern Cooperative Oncology Group(ECOG) ≥ 2
  3. Patients with a surgery experience due to a neoplasm in the stomach.
  4. Patients with complications due to gastric cancer (acute hemorrhage, gastric outlet obstruction or perforation)
  5. Patients with distant metastases (M1) including distant lymph nodes (Retropancreatic, para-aortic, periportal, retroperitoneal, or mesenteric lymph nodes)
  6. Patients without distant metastases but who are, according to a surgeon's judgment, unqualified for radical gastrectomy because of invasions to adjacent organs (T4b).
  7. In the case of localized conglomerated metastatic lymph nodes
  8. Patients who received surgery or radiation therapy for a primary cancer developed in another organ or those with active/synchronous double cancer in recent 5 years.
  9. Patients who participated in another clinical trial or was administered with a different investigational drug in 30 days prior to randomization.
  10. Patients who had any of the following in 6 months before the trial recruitment: myocardial infarction, severe/unstable angina pectoris, coronary/peripheral artery bypass surgery, NYHA class III or IV congestive heart failure, stroke or transient ischemic attack.
  11. Patients with a previous experience of uncontrolled seizure, central nervous system or psychological disorders whose conditions are clinically significant to the extent that they are unable to express consent to participate in the trial and oral drug administration is not possible.
  12. Patients with uncontrolled active infection or sepsis.
  13. Patients who had deep vein thrombosis in recent 4 weeks before the beginning of the trial recruitment.
  14. Patients with serious acute or chronic disease that can degrade the patient's ability to participate in the trial or impede the interpretation of the trial results.
  15. Pregnant or breast-feeding patients. Fertile female patients who are positive in pregnancy test.

      Drug Administration for Neoadjuvant Chemotherapy
  16. Inadequate functions of marrow or organs:

      I. Absolute Neutrophil Count (ANC) < 1.5 x 109/L II. Platelet (PLT) < 100 x 109/L III. Hemoglobin (Hb) ≤ 9 g/dL IV. AST> 2.5 x ULN, ALT> 2.5 x ULN V. ALP > 2.5 x ULN VI. Total Bilirubin (T. Bil) > 1.5 x ULN VII. Serum creatinine (Cr) > 1.5 x ULN
  17. Patients who have peripheral neuropathy with clinical signs of Grade≥2 (NCI CTCAE v4.03) or with absence of deep tension reflex (DTR).
  18. Patients with hypersensitivity history of the investigational drug (5-FU, Oxaliplatin, Docetaxel).
  19. Patients who are on treatment with warfarin or coumarin anticoagulants.
  20. Patients who are on immunosuppressive therapy.
  21. Patients who are receiving co-medication with Cytochrome P450 2A6 inducer, inhibitor, and substrate.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 238 (Estimated)
Dates: Start 2021-01 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Number of harvested lymph nodes in D2 lymph node dissection | 2 weeks after operation when the pathologic report is available
  number of lymph nodes, pathologically proven after surgery

SECONDARY OUTCOMES:
3 year progression free survival | 3 years after randomization
  PFS is defined as time from the point of randomization to objective tumor progression or relapse, or to death according to RECIST 1.1.
3 year relapse free survival | 3 years after randomization
  RFS is defined as time from the point of randomization to tumor relapse or death
Comparison of postoperative morbidity and mortality | 90 days after operation
  Defined as the incidence of complications within 30 days after surgery, death rate within 90 days. Classification and severity of the complications shall be based on that of KLASS-02-RCT.
Curative resection rate | 2 weeks after operation when the pathologic report is available
  Defined as a case where complete removal of all tumors were confirmed through gross or microscopic examination; negative resection margin was obtained; and, D2 lymph node dissection was performed.
Conversion to open surgery | 1 day
  Defined as a case which the laparoscopic surgery was converted to an open surgery in the operation time, because of reasons including combined organ resection due to adjacent organ invasion, severe intra-abdominal adhesion, or serious intraoperative bleeding.

IPD SHARING:
Plan to Share IPD: No